CLINICAL TRIAL: NCT03850730
Title: An Open-label, Non-randomized Study of the Efficacy of Pazopanib for the Treatment of Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Pazopanib for the Treatment of Epistaxis in Hereditary Hemorrhagic Telangiectasia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cure HHT (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HT3
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Epistaxis
Keywords: osler-weber-rendu; nose bleeds; open label; HHT; Pazopanib
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — pazopanib

STUDY DESIGN:
Intervention Model Description: After at least a 6 week baseline, patients will be placed on very low dose Pazopanib [25mg-similar], for 8 weeks.. If the primary bleeding duration endpoint is achieved, than the patient will continue for another 8wks, or a total of 16 weeks on the same dose. Lack of any response will result in a dose advance to 50mg for another 3mths. If a moderate change has occurred, than the 25mg dose will be continued for another 4 weeks, and if primary endpoint achieved, continue for another 12 weeks... Lack of endpoint achievement, will augment dose to 50mg and extend study for 12 weeks, or a total of 24 weeks.
Masking Description: This is an open label study and thus all personnel and patients will be aware of the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pazopanib (Experimental): Pazopanib, initiated after a baseline period at 25mg oral dosing daily, for this one treatment arm, to be compared to the patient's baseline. If endpoint not achieved and safety demonstrated in 2-3mths, an advance of dose to 50mg daily for the ensuing 3mths of study will be considered.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Active pharmaceutical ingredient plus excipients filled into a capsule for the lower dosing necessary in this study
  Other Names: Pazopanib capsule

SUMMARY:
Investigators will test the value of very low dose Pazopanib administered to patients with hereditary hemorrhagic telangiectasia for the reduction in the severity of nose bleeds in those with frequent and long duration bleeding episodes.

DETAILED DESCRIPTION:
Based on frequency and nose bleed duration, a non-randomized, single arm, open label study of 30 hereditary hemorrhagic telangiectasia patients will be treated with very low dose Pazopanib [25mg-similar] for between 16 and 24 weeks.. The primary endpoint is a reduction in bleeding duration of 50% or more, along with multiple secondary related endpoints, including bleed frequency, blood counts and quality of life; as compared to 6-12 weeks of baseline characteristics. If after the first 8 weeks of therapy benefit is suboptimal, dose advance to 50mg-similar daily can be considered.

ELIGIBILITY:
Inclusion Criteria:

* a definite diagnosis of hereditary hemorrhagic telangiectasia defined as having at least 3 of the following criteria:

  * Spontaneous and recurrent epistaxis.
  * Multiple telangiectasias at characteristic sites: lips, oral cavity, fingers, nose.
  * Visceral lesions: GI telangiectasia, pulmonary, hepatic, cerebral or spinal AVMs.
  * A first degree relative with hereditary hemorrhagic telangiectasia according to these criteria.
  * OR a gene sequencing diagnosis of hereditary hemorrhagic telangiectasia

    2. Epistaxis due to hereditary hemorrhagic telangiectasia at least 2x per week, for a cumulative duration of at least 25 minutes per week

    3. Epistaxis is clinically stable during the 12 weeks prior to screening in the clinical judgment of the investigator (i.e. no major changes in frequency or duration of epistaxis).

    4. Participant agrees not to undergo cautery of nasal telangiectasias or take any experimental therapies for hereditary hemorrhagic telangiectasia other than the study drug while participating in the study.

    5. Male or female [non-child bearing potential]

Exclusion Criteria:

1. Participant has known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib that in the opinion of the investigator contradicts their participation.
2. Currently has untreated cerebral arterio-venous malformations (AVMs), cerebral arteriovenous fistulae, or cerebral cavernous malformations (CCMs) (Note: MRI scan does not need to be repeated at screening if AVMs, arterio-venous fistulas and CCMs were absent on a scan at age ≥18 years).
3. Currently has perfused pulmonary AVMs with feeding artery diameter >3mm.
4. Known significant bleeding sources other than nasal or gastrointestinal.
5. Systemic use of a vascular endothelial growth factor inhibitor in the past 3 months or previous enrollment in this study.
6. Active and recent onset of clinically significant diarrhea.
7. Current or recent (in the last 5 years) malignancies (except non-melanoma skin cancers)
8. Participant has had major surgery (e.g. surgical ligation of an AVM) or trauma within 28 days or had minor surgical procedures (e.g. central venous access line removal) within 7 days prior to dosing, the latter representing a recent wound, fracture or ulcer
9. Participant has a planned surgery during the period to include active treatment and 6 weeks of follow up.
10. Participant has clinically significant gastrointestinal abnormalities (other than hereditary hemorrhagic telangiectasia related vascular lesions)
11. Participant during the 6 months prior to first dose of study drug has a history of cerebrovascular accident (including transient ischemic attacks), pulmonary embolism, untreated deep vein thrombosis (DVT), myocardial infarction, or any other thrombotic event.
12. QTc ≥450 msec, based on averaged QTc values of triplicate ECGs obtained over a brief recording period [The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual overread. The same QT correction formula must be used for each individual participant to determine eligibility for and withdrawal from the study.]
13. Hgb <6 g/dL.
14. Platelets < 100x109/L.
15. International normalized ratio (INR) >1.2x upper limit of normal and activated partial thromboplastin time (aPTT)>1.2x upper limit of normal.
16. Alanine Transaminase >2x upper limit of normal.
17. Bilirubin >1.5x upper limit of normal (isolated bilirubin >1.5x upper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin <35%).
18. Participant has poorly controlled hypertension [defined as systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥90 mmHg. Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry [between screen and baseline]. At Screening, blood pressure must be assessed three times and the mean SBP/DBP must be <140/90 mmHg in order for a participant to be eligible for the study.]
19. Substantive renal disease (eGFR <30 mL/min/1.73m2calculated using the Cockcroft-Gault formula)
20. Echo derived left ventricular ejection fraction <30%.
21. Thyroid stimulating hormone > upper limit of normal.
22. Urine protein to creatinine ratio >0.3.
23. Neutrophil count <1500/mm3.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in epistaxis duration in minutes | Summed minutes of bleeding at baseline 3 weeks and the last 3 weeks of dosing, over16-24 weeks of dosing
  A daily electronic record of each bleed, with start and end time, provides the daily epistaxis duration, compounded over each 3 weeks of study time

SECONDARY OUTCOMES:
Percent change in average gushing frequency | Last 3 weeks of drug period vs baseline 3 weeks; over 16-24 weeks of dosing
  Patient rated intensity of each bleed, as in 0 or 1, averaged over 3 wk periods.
Percent change in average bleed frequency | Last 3 weeks compared to the baseline 3 weeks; over 16-24 weeks of dosing
  Annotated number of bleeds per day, and summed over 3 week periods
Absolute [gm/dl] change in serum hemoglobin | comparing last 6 weeks to baseline 3-6 weeks; over 16-24 weeks of drug dosing
  Serum values drawn every 3 weeks
Change in the frequency of blood transfusions | Final 6 weeks of study, compared to baseline 3-6 weeks; over 16- 24 weeks of dosing
  Use of packed red blood cells over 6 week time periods.
Change in the frequency of IV iron infusions | Last 6 weeks of dosing to first 6 weeks; over 16-24 weeks of drug administration
  Number of interval IV iron infusions in 6 week periods
Percent change in the per bleed average epistaxis severity | The final 3 weeks to the baseline 3 weeks of the study; for a16-24 week duration study
  Epistaxis severity score [0-10] housed in the current patient reported outcome instrument will be averaged
Daily monitoring for change in systolic blood pressure [mm mercury] using daily recordings | Daily from baseline through up to 24 weeks till on-drug study completion.
  Patients rising above 140 mm mercury, or those who increase by 20 or more mm mercury will trigger protocol defined treatments.
Daily monitoring for change in diastolic blood pressure [mm mercury] | Daily from baseline through up to 24 weeks till on-drug study completion
  Patients rising above 90 mm mercury, or those who increase by 10 mm mercury or more will trigger protocol defined treatments.
Number of participants with changes in alanine aminotransferase [liver function test] | Baseline and throughout the 16-24 week dosing period
  measurement every 3 weeks to evaluate fold increase with use of drug
Monitor for active and safe trough serum drug concentrations | Over 16-24 week duration of study; once at steady state for each administered dose
  Assays to be analyzed to evaluate the exposures done to remain within safe and effective range [1ug/ ml to 10ug/ml].....
Evaluate for change in composite mental quality of life scores | baseline, week 12 and at study drug-dosing end; 16, 20 or 24weeks
  short form health survey 36 [range 1-100, higher number representing better self-reported mental health]
Evaluate for change in composite physical quality of life scores | baseline, week 12 and at study drug-dosing end; up to 24 weeks.
  short form health survey 36 [range 1-100, higher number representing better self-reported physical health]
Evaluate for change in fatigue composite scores | baseline and study end; up to 24 weeks
  Patient-report outcome measurement information system-fatigue; [0-100 scale; lower number representing less fatigue]. Queries the degree of fatigue and the implications on physical functioning. Reduction of 5 or more in the composite score represents clinically relevant reductions in fatigue.

OTHER OUTCOMES:
Interrogate levels of Iron stores | baseline and at on-drug study end; 16, 20 or 24 weeks depending on study duration
  Ferritin serum levels [normal range 12 ug/ ml to 150ug/ml female, 300ug/ ml male]. However, above 30ug/ ml valued as relevant for proper erythropoiesis]
Characterize change in left ventricular stress | baseline and on-drug study end; 16, 20 or 24 weeks depending on study duration]
  NTproBNP serum values represent a surrogate for left ventricular stress [<125pg/ml normal, while above 350pg/ml high and potentially consistent with heart failure]

CONTACTS AND LOCATIONS:
Overall Officials: Raj Kasthuri, MD, Principal Investigator — University of North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
After the PI and associates produce the primary and adjunct reports, these data can be posted on data files for public access